CLINICAL TRIAL: NCT03495752
Title: The Effect of Cardiovascular Fatigue on Performance of the Forward-Step-Down Test
Brief Title: The Effect of Fatigue on the Forward-Step-Down Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Erin N. McCallister, Instructor, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00000949
Record Dates: First submitted 2018-04-04; First posted 2018-04-12 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Fatigue
Keywords: muscle performance; injury prevention; step down; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre/Post Repeated Measures (Experimental): Performance on the forward-step-down test (FSDT) before and at one, five, and ten minutes following the Bruce Fatigue Protocol
  Interventions: Other: Bruce Fatigue Protocol

INTERVENTIONS:
Other: Bruce Fatigue Protocol — Participant will perform the Bruce protocol as a fatigue stimulus to examine the impact of fatigue on the FSDT

SUMMARY:
This study investigates the effect that performing a cardiovascular maximum effort test (the Bruce treadmill protocol) has on performance of the Forward-Step-Down Test (FSDT). The FSDT is performed prior to the fatigue protocol as a baseline measurement, then at 1, 5, and 10 minutes after the fatigue protocol. Participants much reach a certain heart rate (within 10 bpm) of their age predicted maximum heart rate to ensure that the fatigue protocol reaches a maximum fatiguing effort.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects that a volitional maximal cardiovascular exertion test (the Bruce Treadmill Protocol) has on performance of the Forward-Step-Down (FSD) test, and to investigate how performance on the FSD test changes at multiple time points following the fatigue test.

Our hypotheses for this study are as follows:

* Null (H0): Participants will not demonstrate a change in score on the FSD test after performance of the Bruce test at any time point.
* Alternate (H1): Participants will demonstrate a change in score on the FSD test after performance of the Bruce test at one or multiple of the repeated measurements.

The FSD test has been shown to correlate with movement quality. Deficits in strength and flexibility that result in movement impairments are associated with scores on the test delineating "moderate" movement quality. Fatigue may play a role in increased injury risk, with fatigued participants in numerous studies showing compromised movement patterns that increase risk of injury. At this time, many of the screening tools used to determine the impact of fatigue on a player's ability to continue to play/practice involved dynamic or explosive movements, and rely on indicators such as femoral internal rotation or hip adduction angles at initial contact to grade movement patterns. These biomechanical indicators may be difficult for non-professional personnel to observe, limiting their use outside a clinic. There is currently no research on the role of the FSD test in assessing for changes in movement pattern that result from fatigue.

The literature currently acknowledges that fatigue results in altered movement patterns. Several studies have investigated the impact that fatigue has on performing challenging movements, such as plyometric drop jumps, cutting, jumping and running, and landing. However, with higher level assessments such as these, there is an increased risk for injury if performed while fatigued. Therefore, a lower level test, such as the FSD test, would be ideal as a safe and effective screening tool to look at the impact of fatigue stimulus (game play) on a person's movement quality. As stated above, the FSD test has been validated as a measure of movement quality, with acceptable interrater reliability. In addition, poor movement quality during the FSD test has been shown to correlate with several impairments such as hip abductor strength and poor flexibility. Existing literature discusses the impact of the hip abductors on knee position and risk for knee injury. Therefore, a functional test that assesses not only movement quality but identifies possible causes of poor movement would be ideal for preventing injury. Research has shown difference in postural balance following aerobic fatigue depending on the time since fatigue, with poor performance immediately following but improved performance 10 minutes after the fatigue stimulus was stopped. Therefore, this study will examine the FSD test at one, five, and ten minutes following the cardiovascular fatigue protocol in order to discern performance differences in movement quality related to time/recovery. These differences may be important because if the FSD test can be used as a screening tool to examine a person's fatigue level, it is important to also know the appropriate time to use the test in order to get accurate results.

In this study, the Bruce test is used to achieve cardiovascular fatigue. Clinically it is a "VO2max" (maximum volume of oxygen consumption) prediction test and is intended to continue to the point of failure (maximum test). In a true VO2max test, the participant performs the cardiovascular test until respiratory spirometry measures a plateau of the VO2, or oxygen consumption, between two workloads. This is indicative of that participant's maximum cardiovascular physiological limits. During a true VO2max test, respiratory gases are analyzed as well as heart rate, blood pressure, and sometimes blood lactate samples are obtained. Together these values determine the success in reaching a true VO2max test, demonstrate cardiovascular fatigue, and ensure safety of the participant. Often, this point is not reached in untrained or unhealthy individuals.

Performing a true VO2max test is more expensive and time-consuming for the participant than performing a maximal or submaximal graded exercise test. Therefore, the Bruce protocol uses mathematical derivation to predict VO2max from the participant's performance on the Bruce. To estimate an accurate prediction of the VO2max and ensure cardiovascular fatigue, the target heart rate is often set at within 10 bpm of the age-predicted maximum heart rate when using a lower error formula such as the Tanaka formula. Therefore, in this study participants' age-predicted maximum heart rate will be calculated using the formula derived by Tanaka with an acceptable variability of within 10 bpm at the maximum heart rate measured during the Bruce. The Tanaka formula is accurate for a population of healthy men and women. In this study, "healthy" is defined as being in the "low risk" category for exercise as stated by the American College of Sports Medicine, and is one of the inclusion criteria for this study.

* Prior to performing the testing, participants will be consented and screened for inclusion and exclusion criteria at the end of an exercise physiology class during the summer 2018 semester. This will occur before the students begin their exercise testing labs in which the Bruce protocol is performed. Following consenting, participants will proceed to the testing during the four-week data collection period during the summer 2018 semester.
* Each participant will perform the pre-and post-testing in the same day. The pre-fatigue FSD test occurs just prior to the fatigue (Bruce) protocol, and the post-testing will occur at one, five, and ten minutes after completion of the fatigue protocol. Initial resting heart rate will be measured, as will heart rate at 0, 30, and 60 seconds following completion of the Bruce to ensure appropriate heart rate responses to exercise for a healthy young adult as per the inclusion criteria of participants being "low risk" for adverse events during vigorous exercise.
* The expected duration to obtain all necessary participants is up to 4 weeks.
* The estimated time for the researches to perform the primary analysis is 3 months
* The estimated time to prepare the manuscript for publication is 1 year.

This study will be a repeated-measures design, with all participants undergoing both pre- and post-fatigue FSD test assessments. Two orthopaedic specialist physical therapists will perform the FSD assessments. The investigators will review scoring guidelines per the Park article, and will practice scoring the test prior to data collection to ensure good interrater reliability. Scores on the FSD test from each assessor will be averaged after data collection and prior to data analysis, with each assessor blinded to the other's score prior to averaging the scores. Participants will be healthy physical therapy students. Fatigue will be induced via the Bruce protocol used in assessment of maximum cardiovascular capacity. The treadmill used is an HP Cosmos Quasar (HP Cosmos, Germany). The heart rate monitors used are Polar monitors (Polar Electro Inc, Bethpage, NY)

The FSD test grades the participant on movement quality during a repeated step down from a 20 cm step. The weight bearing leg will be the dominant leg (the leg the participant would use to kick a ball) as used in the Park et al experiment. The FSD test consists of five repeated movements of the forward step down, with one score given for the whole set of five repetitions. For each set of five movements, the rater observes and produces one score for that set of five movements. For data analysis, the investigators will use the average of each score for each FSD test. For example, on the pre-test for a participant, if one investigator scored the pre-test FSD a 2/6, and the second investigator scored the pre-test a 1/6, the "averaged" score for the participant's pre-test is a 1.5/6. This same procedure would be repeated for the three post-test FSD tests.

The Bruce protocol is self-limited with participants stopping at maximal exertion. Maximal exertion will be defined as within 10 bpm of the participants predicted maximum heartrate as calculated by the formula "208-(0.7 x age)" derived by Tanaka from a population of healthy men and women. The within 10 bpm heart rate cutoff has been used as a benchmark of achieving maximal exertion in a maximal exercise test based off the calculated maximum heart rate using the Tanaka formula. The participants' Borg Rating of Perceived Exertion (RPE) will also be recorded as part of the Bruce protocol; however, since the participants know they will have to perform the FSD test following the Bruce protocol, the investigators will use heart rate instead of RPE as a metric for exertion due to its more objective nature and to avoid a possible threat to validity of the fatigue protocol. During the Bruce protocol, treadmill speed and incline are increased every three minutes until the subject volitionally stops the test at maximal exertion. Heart rate and RPE are monitored each minute during the Bruce protocol, with assessment of blood pressure prior and following the treadmill test as part of the Exercise Physiology class.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited from current physical therapy students in the class of 2020 who are enrolled in PHTH 7565. During the consent process, the participants will be screened using the American College of Sports Medicine's guidelines for safe participation in vigorous exercise. By meeting the ACSM criteria, the participant is considered low risk for adverse events while participating in vigorous activity. Finally, in order for the student to participate, they must achieve within 10 bpm of their predicted maximum heart rate, as calculated by the Tanaka formula as stated above.

Exclusion Criteria:

* 3.2 Exclusion criteria are pre-existing cardiovascular conditions or diseases that prevent participation in a maximal effort test without physician clearance per the ACSM guidelines. Participants who do not reach their calculated target heart rate by the end of the Bruce protocol will be withdrawn from the study and will not complete post-fatigue testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Change in Score on the Forward-Step-Down Test | up to 10 minutes after intervention
  The participants' scores on the pre-test FSDT will be compared to their scores post-test measured at 1, 5, and 10 minutes after the fatigue stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Erin McCallister, DPT, Principal Investigator — LSUHSC-Shreveport
Locations (1):
- LSUHSC-Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park KM, Cynn HS, Choung SD. Musculoskeletal predictors of movement quality for the forward step-down test in asymptomatic women. J Orthop Sports Phys Ther. 2013;43(7):504-10. doi: 10.2519/jospt.2013.4073. Epub 2013 Jun 11. PMID 23756380
- [Background] Cortes N, Greska E, Kollock R, Ambegaonkar J, Onate JA. Changes in lower extremity biomechanics due to a short-term fatigue protocol. J Athl Train. 2013 May-Jun;48(3):306-13. doi: 10.4085/1062-6050-48.2.03. Epub 2013 Feb 20. PMID 23675789
- [Background] Geiser CF, O'Connor KM, Earl JE. Effects of isolated hip abductor fatigue on frontal plane knee mechanics. Med Sci Sports Exerc. 2010 Mar;42(3):535-45. doi: 10.1249/MSS.0b013e3181b7b227. PMID 19952814
- [Background] Johnston RB 3rd, Howard ME, Cawley PW, Losse GM. Effect of lower extremity muscular fatigue on motor control performance. Med Sci Sports Exerc. 1998 Dec;30(12):1703-7. doi: 10.1097/00005768-199812000-00008. PMID 9861603
- [Background] McLean SG, Samorezov JE. Fatigue-induced ACL injury risk stems from a degradation in central control. Med Sci Sports Exerc. 2009 Aug;41(8):1661-72. doi: 10.1249/MSS.0b013e31819ca07b. PMID 19568192
- [Background] Mohammadi F, Roozdar A. Effects of fatigue due to contraction of evertor muscles on the ankle joint position sense in male soccer players. Am J Sports Med. 2010 Apr;38(4):824-8. doi: 10.1177/0363546509354056. Epub 2010 Feb 5. PMID 20139329
- [Background] Wesley CA, Aronson PA, Docherty CL. Lower Extremity Landing Biomechanics in Both Sexes After a Functional Exercise Protocol. J Athl Train. 2015 Sep;50(9):914-20. doi: 10.4085/1062-6050-50.8.03. Epub 2015 Aug 18. PMID 26285090
- [Background] Moran KA, Clarke M, Reilly F, Wallace ES, Brabazon D, Marshall B. Does endurance fatigue increase the risk of injury when performing drop jumps? J Strength Cond Res. 2009 Aug;23(5):1448-55. doi: 10.1519/JSC.0b013e3181a4e9fa. PMID 19620920
- [Background] Padulo J, Attene G, Ardigo LP, Bragazzi NL, Maffulli N, Zagatto AM, Dello Iacono A. Can a Repeated Sprint Ability Test Help Clear a Previously Injured Soccer Player for Fully Functional Return to Activity? A Pilot Study. Clin J Sport Med. 2017 Jul;27(4):361-368. doi: 10.1097/JSM.0000000000000368. PMID 27428681
- [Background] Ros AG, Holm SE, Friden C, Heijne AI. Responsiveness of the one-leg hop test and the square hop test to fatiguing intermittent aerobic work and subsequent recovery. J Strength Cond Res. 2013 Apr;27(4):988-94. doi: 10.1519/JSC.0b013e31825feb5b. PMID 22706574
- [Background] Herman G, Nakdimon O, Levinger P, Springer S. Agreement of an Evaluation of the Forward-Step-Down Test by a Broad Cohort of Clinicians With That of an Expert Panel. J Sport Rehabil. 2016 Aug;25(3):227-32. doi: 10.1123/jsr.2014-0319. Epub 2015 Dec 14. PMID 26655963
- [Background] Steinberg N, Eliakim A, Zaav A, Pantanowitz M, Halumi M, Eisenstein T, Meckel Y, Nemet D. Postural Balance Following Aerobic Fatigue Tests: A Longitudinal Study Among Young Athletes. J Mot Behav. 2016 Jul-Aug;48(4):332-40. doi: 10.1080/00222895.2015.1095153. Epub 2016 Jan 5. PMID 26731202
- [Background] ACSM's Guidelines for Exercise Testing and Prescription. 10 ed. Philadelphia, PA: Wolters Kluwer; 2018.
- [Background] Beltz NM, Gibson AL, Janot JM, Kravitz L, Mermier CM, Dalleck LC. Graded Exercise Testing Protocols for the Determination of VO2max: Historical Perspectives, Progress, and Future Considerations. J Sports Med (Hindawi Publ Corp). 2016;2016:3968393. doi: 10.1155/2016/3968393. Epub 2016 Dec 25. PMID 28116349
- [Background] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730
- [Background] Riebe D, Franklin BA, Thompson PD, Garber CE, Whitfield GP, Magal M, Pescatello LS. Updating ACSM's Recommendations for Exercise Preparticipation Health Screening. Med Sci Sports Exerc. 2015 Nov;47(11):2473-9. doi: 10.1249/MSS.0000000000000664. PMID 26473759

DOCUMENTS (1):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT03495752/Prot_000.pdf